CLINICAL TRIAL: NCT02440854
Title: A Multicentre, Cohort Study to Assess the Impact on SYMptom Burden and Patient Health-related Quality of Life of Afatinib Treatment in Advanced Non-small Cell Lung Cancer in a Real World Setting in Greece.
Brief Title: Evaluate the Impact of Afatinib on Quality of Life and Symptom Burden of Greek Subjects With Advanced NSCLC in Routine Patient Care Settings
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200.247
Record Dates: First submitted 2015-04-28; First posted 2015-05-12 (Estimated); Results first posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with non-small cell lung cancer (NSCLC) treated with afatinib: Patients with advanced/metastatic non-small cell lung cancer (NSCLC) in Greece treated with afatinib. Patients were treated as per the routine medical practice in terms of visit frequency, types of assessments performed and with adherence to the local prescribing requirements for afatinib. Patients were observed in the context of the study until the end of study participation, defined as a maximum of 48 months after afatinib treatment initiation or until disease progression, death, withdrawal of consent, unacceptable toxicity, study completion or physician's decision whichever occurred earlier.
  Interventions: Drug: afatinib

INTERVENTIONS:
Drug: afatinib — Patients were treated as per the routine medical practice in terms of visit frequency, types of assessments performed and with adherence to the local prescribing requirements for afatinib.

SUMMARY:
This non-interventional study will include a representative sample of patients with locally advanced or metastatic NSCLC harboring Epidermal Growth Factor Receptor (EGFR)-mutations in Greece. Eligible NSCLC patients, for whom the physician has decided to initiate treatment with the study medication (afatinib, GIOTRIF®) will be treated according to the local prescribing information and standard medical practice in terms of visit frequency and types of assessments performed.

The study will investigate the impact of GIOTRIF (Afatinib) on patients' disease-related symptom burden and Health-Related Quality of Life (HRQoL) in a real world clinical setting in Greece.The Average Symptom Burden Index (ASBI) score of the Lung Cancer Symptom Scale (LCSS) in eligible patients, after 6 months of therapy, will be analyzed.

The overall study duration period is expected to be 60 months, including a 48-month enrollment period and a minimum 12-month follow-up period.

DETAILED DESCRIPTION:
Study Design:

ELIGIBILITY:
Inclusion criteria:

* Adult outpatients (18 years and older) of either gender;
* Histologically or cytologically confirmed locally advanced or metastatic (IIIB/IV) NSCLC of any histological type with activating EGFR mutation(s) according to local laboratory EGFR testing;
* EGFR- tyrosine kinase inhibitor (TKI) naive patients;
* Patients for whom the decision to prescribe therapy with afatinib (GIOTRIF®) according to the locally approved product's summary of product characteristics (SmPC) has already been taken prior to their enrolment in the study; the assignment of the patient to this therapeutic strategy is not decided in advance by the study protocol but falls within current practice and the prescription of afatinib is clearly separated from the physicians decision to include the patient in the current study;
* Patients must be able and willing to provide written informed consent and to comply with the requirements of this study protocol;

Exclusion criteria:

* Patients who have initiated treatment with Afatinib more than 7 days prior to their enrolment into the study;
* Patients that meet any of the contraindications to the administration of the study drug according to the approved SmPC;
* Receipt of any investigational agent within 30 days or 5 half-lives of the investigational agent (whichever is longer) before the commencement of therapy with afatinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: NSCLC EGFR mutation
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2021-02-17 (Actual); Study Completion 2021-02-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (7):
- Greece (7):
  - University General Hospital of Evros, Alexandroupoli
  - Chest Hospital of Athens "Sotiria", Athens
  - "Attikon" University General Hospital of Attica, Haidari
  - University General Hospital of Heraklion, Heraklion
  - Bioclinic Thessaloniki, Thessaloniki
  - Interbalkan Medical Center of Thessaloniki, Thessaloniki
  - General Hospital of Thessaloniki "G. Papanikolaou", Thessaloniki

REFERENCES:
- See also: Related Info — https://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a non-interventional, multicentre, cohort study, based on new data collection, which included a representative sample of patients with advanced/metastatic Non-small cell lung cancer (NSCLC) in Greece.
Pre-assignment Details: Patients were treated according to the local prescribing information of the study medication (afatinib, GIOTRIF®) and routine medical practice in terms of visit frequency and types of assessments performed. The assignment of the patient to this therapeutic strategy was not decided in advance by the study protocol but fell within current practice and the prescription of afatinib was clearly separated from the physician's decision to include the patient in the current study.
Period: Overall Study
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Started (Enrolled) | 80
Analyzed | 77
Completed (Completed 48 month follow up) | 0
Not Completed | 80
Not completed — Relocation of patient | 1
Not completed — Death | 6
Not completed — Lost to Follow-up | 10
Not completed — Afatinib discontinuation | 46
Not completed — stopped study at earlier timepoint | 14
Not completed — Study medication not received | 1
Not completed — Violation of inclusion criteria | 2

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): all eligible subjects that have received at least one dose of afatinib in the study.
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 77
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 77
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Experienced a Minimum Clinically Important Improvement in Symptoms Over 6 Months of Treatment
Description: Number of patients who experience a minimum clinically important improvement in symptoms is reported. A patient was categorized as having an improvement if the mean score of any two consecutive post-baseline Average Symptom Burden Index (ASBI) score of Lung Cancer Symptom Scale (LCSS) assessments for that patient was at least 10 points below the patient's ASBI score of LCSS at enrolment, over 6 months of treatment.
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Each item is scored on a 100-millimeter (mm) Visual Analogue Scale (VAS), with score reported from 0 to 100, with 0 representing the best score. ASBI score was calculated by the mean of the 6 major lung cancer symptoms (loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis). For a given assessment, if any of the six symptom-specific questions was not completed, the ASBI score was not calculated.
Time Frame: Baseline and 6 months following start of treatment.
Population: All eligible subjects that have received at least one dose of afatinib in the study and who had two consecutive post-baseline Lung Cancer Symptom Scale (LCSS) Average Symptom Burden Index (ASBI) assessments over the 6-month treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 53
Participants | 13

2. Secondary Outcome: Patient-rated Average Symptom Burden Index (ASBI) Score of Lung Cancer Symptom Scale (LCSS)
Description: Patient-rated ASBI score of LCSS at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study) is reported.
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Each item was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score. ASBI score was calculated by the mean of the 6 major lung cancer symptoms (loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis). For a given assessment, if any of the six symptom-specific questions had not been completed, the ASBI score was not calculated.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: All eligible subjects who have been enrolled into the study regardless of whether or not they have finally completed their projected participation in the study and who provided data to this endpoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 14.1 (12.2)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 11.5 (10.3)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 9.3 (9.0)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 7.1 (8.3)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 7.6 (7.3)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 7.8 (8.7)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 7.6 (10.5)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 5.3 (6.4)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 6.2 (6.5)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 7.5 (8.1)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 11.5 (6.9)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 1.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p = 0.002, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p = 0.014, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p = 0.246, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p = 0.103, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p = 0.004, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p = 0.012, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p = 0.024, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p = 0.009, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.008, t-test, 2 sided; Paired t-test

3. Secondary Outcome: Patient-rated Total Lung Cancer Symptom Scale (LCSS) Score
Description: Patient-rated total LCSS score -defined as the average of the aggregate score of all 9 items that comprise the LCSS- at enrolment and at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Each item was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score. ASBI score was calculated by the mean of the 6 major lung cancer symptoms (loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis). For a given assessment, if any of the six symptom-specific questions had not been completed, the ASBI score was not calculated.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 17.0 (13.1)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 14.7 (11.3)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 12.4 (10.1)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 10.7 (9.2)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 11.7 (8.6)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 11.1 (9.3)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 10.6 (10.6)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 8.3 (7.8)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 9.6 (7.7)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 10.8 (8.8)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 13.8 (7.1)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 4.6 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p = 0.027, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p = 0.030, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p = 0.351, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p = 0.143, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p = 0.163, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p = 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p = 0.003, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p = 0.036, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p = 0.043, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.040, t-test, 2 sided; Paired t-test

4. Secondary Outcome: Patient-rated Lung Cancer Symptom Scale (LCSS) Individual Item Scores: Loss of Appetite
Description: Patient-rated LCSS individual item scores: Loss of appetite at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Loss of appetite was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 17.8 (21.9)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 21.7 (26.2)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 15.9 (19.9)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 14.7 (23.9)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 12.1 (19.4)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 13.6 (22.6)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 11.7 (20.6)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 8.9 (14.8)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 7.4 (7.3)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 7.6 (10.0)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 28.3 (32.2)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p = 0.003, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.163, t-test, 2 sided; Paired t-test

5. Secondary Outcome: Patient-rated Lung Cancer Symptom Scale (LCSS) Individual Item Scores: Fatigue
Description: Patient-rated LCSS individual item scores: Fatigue at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Fatigue was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 27.4 (26.1)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 22.0 (21.8)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 20.3 (18.3)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 16.7 (20.9)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 17.5 (19.9)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 17.2 (17.5)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 14.5 (17.1)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 12.6 (16.5)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 14.3 (15.8)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 12.4 (12.1)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 25.1 (20.3)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 6.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p = 0.003, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p = 0.009, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p = 0.012, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p = 0.332, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p = 0.029, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p = 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p = 0.177, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p = 0.436, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p = 0.302, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.291, t-test, 2 sided; Paired t-test

6. Secondary Outcome: Patient-rated Lung Cancer Symptom Scale (LCSS) Individual Item Scores: Cough
Description: Patient-rated LCSS individual item scores: Cough at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Cough was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 14.9 (21.5)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 6.7 (10.9)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 8.5 (14.5)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 4.2 (8.1)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 4.1 (7.5)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 4.1 (8.1)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 6.5 (13.5)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 2.4 (6.1)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 4.0 (6.6)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 10.2 (12.2)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 5.1 (7.6)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p = 0.002, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.025, t-test, 2 sided; Paired t-test

7. Secondary Outcome: Patient-rated Lung Cancer Symptom Scale (LCSS) Individual Item Scores: Dyspnoea
Description: Patient-rated LCSS individual item scores: Dyspnoea at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Dyspnoea was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 10.8 (17.4)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 7.5 (16.5)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 5.5 (11.6)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 3.4 (8.4)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 3.3 (7.9)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 4.4 (9.1)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 5.2 (13.7)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 2.3 (4.9)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 3.9 (6.9)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 8.5 (13.4)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 5.9 (10.0)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p = 0.003, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.025, t-test, 2 sided; Paired t-test

8. Secondary Outcome: Patient-rated Lung Cancer Symptom Scale (LCSS) Individual Item Scores: Haemoptysis
Description: Patient-rated LCSS individual item scores: Haemoptysis at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Haemoptysis was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 1.6 (5.0)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 1.3 (6.9)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 1.0 (4.4)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 0.9 (2.5)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 1.4 (3.4)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 1.2 (2.8)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 1.4 (3.3)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 1.4 (6.4)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 0.6 (1.5)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 0.9 (1.5)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 0.4 (1.1)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test

9. Secondary Outcome: Patient-rated Lung Cancer Symptom Scale (LCSS) Individual Item Scores: Pain
Description: Patient-rated LCSS individual item scores: Pain at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Pain was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 12.0 (19.4)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 9.7 (16.3)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 4.5 (8.6)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 3.0 (5.4)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 7.2 (14.2)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 6.5 (11.4)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 6.1 (10.9)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 4.2 (8.7)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 7.2 (14.0)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 5.4 (8.3)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 4.4 (6.9)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.002, t-test, 2 sided; Paired t-test

10. Secondary Outcome: Patient-rated Lung Cancer Symptom Scale (LCSS) Individual Item Scores: Overall Symptomatic Distress
Description: Patient-rated LCSS individual item scores: Overall symptomatic distress at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Overall symptomatic distress was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score. ASBI score was calculated by the mean of the 6 major lung cancer symptoms (loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis). For a given assessment, if any of the six symptom-specific questions had not been completed, the ASBI score was not calculated.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 16.2 (17.7)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 15.9 (15.6)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 17.3 (0.0)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 13.8 (16.3)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 14.8 (16.7)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 12.7 (14.5)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 12.1 (13.4)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 12.0 (12.7)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 11.7 (12.7)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 11.0 (7.3)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 8.6 (7.1)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 10.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p = 0.022, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p = 0.004, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p = 0.032, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p = 0.066, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p = 0.042, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p = 0.045, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p = 0.014, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p = 0.015, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.462, t-test, 2 sided; Paired t-test

11. Secondary Outcome: Patient-rated Lung Cancer Symptom Scale (LCSS) Individual Item Scores: Interference With Normal Activity
Description: Patient-rated LCSS individual item scores: Interference with normal activity at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Interference with normal activity was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score. ASBI score was calculated by the mean of the 6 major lung cancer symptoms (loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis). For a given assessment, if any of the six symptom-specific questions had not been completed, the ASBI score was not calculated.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 22.8 (26.3)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 19.6 (20.8)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 16.7 (17.4)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 16.3 (16.1)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 18.1 (17.9)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 15.9 (16.5)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 16.1 (15.4)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 12.6 (17.4)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 15.5 (12.0)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 17.7 (14.3)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 10.6 (16.9)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 13.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p = 0.004, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p = 0.008, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p = 0.315, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p = 0.237, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p < 0.001, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p = 0.002, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p = 0.004, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p = 0.010, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.683, t-test, 2 sided; Paired t-test

12. Secondary Outcome: Patient-rated Lung Cancer Symptom Scale (LCSS) Individual Item Scores: Global Quality of Life (QoL)
Description: Patient-rated LCSS individual item scores: Global Quality of Life (QoL) at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The patient-rated scale consists of six symptom-specific questions that address loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis. Global Quality of Life (QoL) was scored on a 100-mm Visual Analogue Scale (VAS), with scores reported from 0 to 100 with 0 representing the best score. ASBI score was calculated by the mean of the 6 major lung cancer symptoms (loss of appetite, fatigue, cough, dyspnoea, pain and haemoptysis). For a given assessment, if any of the six symptom-specific questions had not been completed, the ASBI score was not calculated.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
score on a scale
  Baseline | 29.6 (24.8)
  Month 2: number analyzed (Participants) | 55
  Month 2 | 27.8 (23.0)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 23.8 (18.6)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 23.5 (21.8)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 26.9 (23.0)
  Month 10: number analyzed (Participants) | 35
  Month 10 | 24.5 (20.6)
  Month 12: number analyzed (Participants) | 35
  Month 12 | 21.9 (16.0)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 18.2 (16.8)
  Month 24: number analyzed (Participants) | 19
  Month 24 | 22.1 (17.1)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 23.7 (16.0)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 36.1 (34.1)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 12.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p = 0.062, t-test, 2 sided; Paired t-test
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p = 0.062, t-test, 2 sided; Paired t-test
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p = 0.027, t-test, 2 sided; Paired t-test
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p = 0.170, t-test, 2 sided; Paired t-test
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p = 0.271, t-test, 2 sided; Paired t-test
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p = 0.002, t-test, 2 sided; Paired t-test
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p = 0.003, t-test, 2 sided; Paired t-test
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p = 0.157, t-test, 2 sided; Paired t-test
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p = 0.064, t-test, 2 sided; Paired t-test
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.439, t-test, 2 sided; Paired t-test

13. Secondary Outcome: Percentage of Patients With Reported Problems for the European Quality of Life-5 Dimensions-3 Level (EQ-5D-3L) Utility Index Score Dimension: Mobility
Description: Percentage of patients with reported problems for the EQ-5D-3L utility index score dimension: Mobility.
  The EQ-5D-3L descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1="no problems"; 2="some problems"; 3= "extreme problems". Reported are the percentage of patients with problem, consisting of both level 2 ("some problems") and level 3 ("extreme problems") with the remaining subjects having reported level 1 ("no problems").
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
Percentage of patients
  Baseline | 44.7
  Month 2: number analyzed (Participants) | 56
  Month 2 | 30.4
  Month 4: number analyzed (Participants) | 54
  Month 4 | 22.2
  Month 6: number analyzed (Participants) | 47
  Month 6 | 17.0
  Month 8: number analyzed (Participants) | 40
  Month 8 | 35.0
  Month 10: number analyzed (Participants) | 36
  Month 10 | 30.6
  Month 12: number analyzed (Participants) | 38
  Month 12 | 28.9
  Month 18: number analyzed (Participants) | 25
  Month 18 | 28.0
  Month 24: number analyzed (Participants) | 22
  Month 24 | 27.3
  Month 30: number analyzed (Participants) | 10
  Month 30 | 10.0
  Month 36: number analyzed (Participants) | 8
  Month 36 | 25.0
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 2 post-baseline, according to problems/no problems; Test type: Other; p = 0.388, McNemar
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 4 post-baseline, according to problems/no problems; Test type: Other; p = 0.006, McNemar
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 6 post-baseline, according to problems/no problems; Test type: Other; p = 0.077, McNemar
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 8 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 10 post-baseline, according to problems/no problems; Test type: Other; p = 0.508, McNemar
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 12 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 18 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 24 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 30 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 36 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar

14. Secondary Outcome: Percentage of Patients With Reported Problems for the European Quality of Life-5 Dimensions-3 Level (EQ-5D-3L) Utility Index Score Dimension: Self-care
Description: Percentage of patients with reported problems for the EQ-5D-3L utility index score dimension: Self-care.
  The EQ-5D-3L descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1="no problems"; 2="some problems"; 3= "extreme problems". Reported are the percentage of patients with problem, consisting of both level 2 ("some problems") and level 3 ("extreme problems") with the remaining subjects having reported level 1 ("no problems").
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
Percentage of patients
  Baseline | 22.4
  Month 2: number analyzed (Participants) | 56
  Month 2 | 14.3
  Month 4: number analyzed (Participants) | 54
  Month 4 | 16.7
  Month 6: number analyzed (Participants) | 47
  Month 6 | 14.9
  Month 8: number analyzed (Participants) | 40
  Month 8 | 12.5
  Month 10: number analyzed (Participants) | 36
  Month 10 | 8.3
  Month 12: number analyzed (Participants) | 38
  Month 12 | 10.5
  Month 18: number analyzed (Participants) | 25
  Month 18 | 12.0
  Month 24: number analyzed (Participants) | 22
  Month 24 | 13.6
  Month 30: number analyzed (Participants) | 10
  Month 30 | 10.0
  Month 36: number analyzed (Participants) | 8
  Month 36 | 12.5
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 2 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 4 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 6 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 8 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 10 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 12 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 18 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar

15. Secondary Outcome: Percentage of Patients With Reported Problems for theEuropean Quality of Life-5 Dimensions-3 Level (EQ-5D-3L) Utility Index Score Dimension: Usual Activities
Description: Percentage of patients with reported problems for the EQ-5D-3L utility index score dimension: Usual activities.
  The EQ-5D-3L descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1="no problems"; 2="some problems"; 3= "extreme problems". Reported are the percentage of patients with problem, consisting of both level 2 ("some problems") and level 3 ("extreme problems") with the remaining subjects having reported level 1 ("no problems").
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
Percentage of patients
  Baseline | 39.5
  Month 2: number analyzed (Participants) | 56
  Month 2 | 33.9
  Month 4: number analyzed (Participants) | 54
  Month 4 | 29.6
  Month 6: number analyzed (Participants) | 47
  Month 6 | 21.3
  Month 8: number analyzed (Participants) | 40
  Month 8 | 30.0
  Month 10: number analyzed (Participants) | 36
  Month 10 | 27.8
  Month 12: number analyzed (Participants) | 38
  Month 12 | 31.6
  Month 18: number analyzed (Participants) | 25
  Month 18 | 24.0
  Month 24: number analyzed (Participants) | 22
  Month 24 | 13.6
  Month 30: number analyzed (Participants) | 10
  Month 30 | 40.0
  Month 36: number analyzed (Participants) | 8
  Month 36 | 12.5
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 2 post-baseline, according to problems/no problems; Test type: Other; p = 0.774, McNemar
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 4 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 6 post-baseline, according to problems/no problems; Test type: Other; p = 0.607, McNemar
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 8 post-baseline, according to problems/no problems; Test type: Other; p = 0.774, McNemar
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 10 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 12 post-baseline, according to problems/no problems; Test type: Other; p = 0.453, McNemar
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 18 post-baseline, according to problems/no problems; Test type: Other; p = 0.688, McNemar
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 24 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 30 post-baseline, according to problems/no problems; Test type: Other; p = 0.250, McNemar
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 36 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar

16. Secondary Outcome: Percentage of Patients With Reported Problems for the European Quality of Life-5 Dimensions-3 Level (EQ-5D-3L) Utility Index Score Dimension: Pain/Discomfort
Description: Percentage of patients with reported problems for the EQ-5D-3L utility index score dimension: Pain/discomfort.
  The EQ-5D-3L descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1="no problems"; 2="some problems"; 3= "extreme problems". Reported are the percentage of patients with problem, consisting of both level 2 ("some problems") and level 3 ("extreme problems") with the remaining subjects having reported level 1 ("no problems").
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
Percentage of patients
  Baseline | 47.4
  Month 2: number analyzed (Participants) | 56
  Month 2 | 25.0
  Month 4: number analyzed (Participants) | 54
  Month 4 | 16.7
  Month 6: number analyzed (Participants) | 47
  Month 6 | 14.9
  Month 8: number analyzed (Participants) | 40
  Month 8 | 30.0
  Month 10: number analyzed (Participants) | 36
  Month 10 | 25.0
  Month 12: number analyzed (Participants) | 38
  Month 12 | 28.9
  Month 18: number analyzed (Participants) | 25
  Month 18 | 20.0
  Month 24: number analyzed (Participants) | 22
  Month 24 | 22.7
  Month 30: number analyzed (Participants) | 10
  Month 30 | 30.0
  Month 36: number analyzed (Participants) | 8
  Month 36 | 25.0
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 2 post-baseline, according to problems/no problems; Test type: Other; p = 0.077, McNemar
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 4 post-baseline, according to problems/no problems; Test type: Other; p < 0.001, McNemar
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 6 post-baseline, according to problems/no problems; Test type: Other; p = 0.006, McNemar
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 8 post-baseline, according to problems/no problems; Test type: Other; p = 0.344, McNemar
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 10 post-baseline, according to problems/no problems; Test type: Other; p = 0.146, McNemar
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 12 post-baseline, according to problems/no problems; Test type: Other; p = 0.180, McNemar
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 18 post-baseline, according to problems/no problems; Test type: Other; p = 0.289, McNemar
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 24 post-baseline, according to problems/no problems; Test type: Other; p = 0.125, McNemar
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 30 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 36 post-baseline, according to problems/no problems; Test type: Other; p = 0.500, McNemar

17. Secondary Outcome: Percentage of Patients With Reported Problems for the European Quality of Life-5 Dimensions-3 Level (EQ-5D-3L) Utility Index Score Dimension: Anxiety/Depression
Description: Percentage of patients with reported problems for the EQ-5D-3L utility index score dimension: Anxiety/depression.
  The EQ-5D-3L descriptive system consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: 1="no problems"; 2="some problems"; 3= "extreme problems". Reported are the percentage of patients with problem, consisting of both level 2 ("some problems") and level 3 ("extreme problems") with the remaining subjects having reported level 1 ("no problems").
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Number; unit: Percentage of patients
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
Percentage of patients
  Baseline | 51.3
  Month 2: number analyzed (Participants) | 56
  Month 2 | 64.3
  Month 4: number analyzed (Participants) | 54
  Month 4 | 59.3
  Month 6: number analyzed (Participants) | 47
  Month 6 | 53.2
  Month 8: number analyzed (Participants) | 40
  Month 8 | 50.0
  Month 10: number analyzed (Participants) | 36
  Month 10 | 55.6
  Month 12: number analyzed (Participants) | 38
  Month 12 | 47.4
  Month 18: number analyzed (Participants) | 25
  Month 18 | 48.0
  Month 24: number analyzed (Participants) | 22
  Month 24 | 63.6
  Month 30: number analyzed (Participants) | 10
  Month 30 | 50.0
  Month 36: number analyzed (Participants) | 8
  Month 36 | 50.0
  Month 42: number analyzed (Participants) | 1
  Month 42 | 100
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 2 post-baseline, according to problems/no problems; Test type: Other; p = 0.210, McNemar
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 4 post-baseline, according to problems/no problems; Test type: Other; p = 0.263, McNemar
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 6 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 8 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 10 post-baseline, according to problems/no problems; Test type: Other; p = 0.629, McNemar
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 12 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 18 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 24 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 30 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Shift in patient distribution between baseline and Month 36 post-baseline, according to problems/no problems; Test type: Other; p > 0.999, McNemar

18. Secondary Outcome: EQ-VAS Score
Description: EQ-VAS score at enrolment and at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study).
  The EQ-VAS is a visual analogue scale (VAS) that takes values between 100 (best imaginable health) and 0 (worst imaginable health), on which patients provide a global assessment of their health.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 76
Score on a scale
  Baseline | 75.5 (16.7)
  Month 2: number analyzed (Participants) | 56
  Month 2 | 75.4 (15.0)
  Month 4: number analyzed (Participants) | 54
  Month 4 | 77.2 (13.6)
  Month 6: number analyzed (Participants) | 47
  Month 6 | 77.1 (17.6)
  Month 8: number analyzed (Participants) | 40
  Month 8 | 76.3 (18.8)
  Month 10: number analyzed (Participants) | 36
  Month 10 | 76.6 (18.4)
  Month 12: number analyzed (Participants) | 38
  Month 12 | 80.0 (15.1)
  Month 18: number analyzed (Participants) | 25
  Month 18 | 79.0 (17.4)
  Month 24: number analyzed (Participants) | 22
  Month 24 | 78.6 (14.9)
  Month 30: number analyzed (Participants) | 10
  Month 30 | 76.2 (18.4)
  Month 36: number analyzed (Participants) | 8
  Month 36 | 85.4 (6.1)
  Month 42: number analyzed (Participants) | 1
  Month 42 | 85.0 (NA) — Standard deviation could not be calculated with one participant.
Statistical Analysis 1: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 2-month post-baseline; Test type: Other; p = 0.098, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 4-month post-baseline; Test type: Other; p = 0.359, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 6-month post-baseline; Test type: Other; p = 0.393, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 8-month post-baseline; Test type: Other; p = 0.055, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 10-month post-baseline; Test type: Other; p = 0.124, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 12-month post-baseline; Test type: Other; p = 0.376, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 18-month post-baseline; Test type: Other; p = 0.033, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 24-month post-baseline; Test type: Other; p = 0.048, Wilcoxon (Mann-Whitney)
Statistical Analysis 9: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 30-month post-baseline; Test type: Other; p = 0.071, Wilcoxon (Mann-Whitney)
Statistical Analysis 10: Comparison: Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib; Baseline vs 36-month post-baseline; Test type: Other; p = 0.848, Wilcoxon (Mann-Whitney)

19. Secondary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score 0
Description: Percentage of participants with Eastern Cooperative Oncology Group Performance Status (ECOG PS) score 0 at baseline and at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study). ECOG has 6 grades (0-5, where 0 is the best possible score and 5 the worst):
  0 = Fully active, able to carry on all pre-disease performance without restriction.
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours.
  4. = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  5. = Dead.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 77
Percentage of participants
  Baseline | 59.7
  Month 2: number analyzed (Participants) | 63
  Month 2 | 79.4
  Month 4: number analyzed (Participants) | 59
  Month 4 | 83.1
  Month 6: number analyzed (Participants) | 52
  Month 6 | 76.9
  Month 8: number analyzed (Participants) | 48
  Month 8 | 72.9
  Month 10: number analyzed (Participants) | 42
  Month 10 | 73.8
  Month 12: number analyzed (Participants) | 40
  Month 12 | 72.5
  Month 18: number analyzed (Participants) | 26
  Month 18 | 80.8
  Month 24: number analyzed (Participants) | 23
  Month 24 | 69.6
  Month 30: number analyzed (Participants) | 10
  Month 30 | 100
  Month 36: number analyzed (Participants) | 8
  Month 36 | 100
  Month 42: number analyzed (Participants) | 1
  Month 42 | 100

20. Secondary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score 1
Description: Percentage of participants with Eastern Cooperative Oncology Group Performance Status (ECOG PS) score 1 at baseline and at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study). ECOG has 6 grades (0-5, where 0 is the best possible score and 5 the worst):
  0 = Fully active, able to carry on all pre-disease performance without restriction.
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours.
  4. = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  5. = Dead.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 77
Percentage of participants
  Baseline | 28.6
  Month 2: number analyzed (Participants) | 63
  Month 2 | 17.5
  Month 4: number analyzed (Participants) | 59
  Month 4 | 11.9
  Month 6: number analyzed (Participants) | 52
  Month 6 | 21.2
  Month 8: number analyzed (Participants) | 48
  Month 8 | 27.1
  Month 10: number analyzed (Participants) | 42
  Month 10 | 26.2
  Month 12: number analyzed (Participants) | 40
  Month 12 | 25.0
  Month 18: number analyzed (Participants) | 26
  Month 18 | 15.4
  Month 24: number analyzed (Participants) | 23
  Month 24 | 26.1
  Month 30: number analyzed (Participants) | 10
  Month 30 | 0
  Month 36: number analyzed (Participants) | 8
  Month 36 | 0
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0

21. Secondary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score 2
Description: Percentage of participants with Eastern Cooperative Oncology Group Performance Status (ECOG PS) score 2 at baseline and at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study). ECOG has 6 grades (0-5, where 0 is the best possible score and 5 the worst):
  0 = Fully active, able to carry on all pre-disease performance without restriction.
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours.
  4. = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  5. = Dead.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 77
Percentage of participants
  Baseline | 9.1
  Month 2: number analyzed (Participants) | 63
  Month 2 | 3.2
  Month 4: number analyzed (Participants) | 59
  Month 4 | 5.1
  Month 6: number analyzed (Participants) | 52
  Month 6 | 1.9
  Month 8: number analyzed (Participants) | 48
  Month 8 | 0
  Month 10: number analyzed (Participants) | 42
  Month 10 | 0
  Month 12: number analyzed (Participants) | 40
  Month 12 | 2.5
  Month 18: number analyzed (Participants) | 26
  Month 18 | 0
  Month 24: number analyzed (Participants) | 23
  Month 24 | 0
  Month 30: number analyzed (Participants) | 10
  Month 30 | 0
  Month 36: number analyzed (Participants) | 8
  Month 36 | 0
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0

22. Secondary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score 3
Description: Percentage of participants with Eastern Cooperative Oncology Group Performance Status (ECOG PS) score 3 at baseline and at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study). ECOG has 6 grades (0-5, where 0 is the best possible score and 5 the worst):
  0 = Fully active, able to carry on all pre-disease performance without restriction.
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours.
  4. = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  5. = Dead.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 77
Percentage of participants
  Baseline | 1.3
  Month 2: number analyzed (Participants) | 63
  Month 2 | 0
  Month 4: number analyzed (Participants) | 59
  Month 4 | 0
  Month 6: number analyzed (Participants) | 52
  Month 6 | 0
  Month 8: number analyzed (Participants) | 48
  Month 8 | 0
  Month 10: number analyzed (Participants) | 42
  Month 10 | 0
  Month 12: number analyzed (Participants) | 40
  Month 12 | 0
  Month 18: number analyzed (Participants) | 26
  Month 18 | 3.8
  Month 24: number analyzed (Participants) | 23
  Month 24 | 4.3
  Month 30: number analyzed (Participants) | 10
  Month 30 | 0
  Month 36: number analyzed (Participants) | 8
  Month 36 | 0
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0

23. Secondary Outcome: Percentage of Participants With Eastern Cooperative Oncology Group Performance Status (ECOG PS) Score 4
Description: Percentage of participants with Eastern Cooperative Oncology Group Performance Status (ECOG PS) score 4 at baseline and at the post-baseline predefined timepoints (i.e., every 2 months (± 3 weeks) during the first 12 months of therapy and every 6 months (±3 weeks) thereafter until the end of patient's participation in the study). ECOG has 6 grades (0-5, where 0 is the best possible score and 5 the worst):
  0 = Fully active, able to carry on all pre-disease performance without restriction.
  1. = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work.
  2. = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours.
  3. = Capable of only limited selfcare, confined to bed or chair more than 50% of waking hours.
  4. = Completely disabled. Cannot carry on any selfcare. Totally confined to bed or chair.
  5. = Dead.
Time Frame: Baseline (Day 0) and at month 2, 4, 6, 8, 10, 12, 18, 24, 30, 36 and 42 post baseline.
Population: as for outcome 2
Measure: Number; unit: Percentage of participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 77
Percentage of participants
  Baseline | 1.3
  Month 2: number analyzed (Participants) | 63
  Month 2 | 0
  Month 4: number analyzed (Participants) | 59
  Month 4 | 0
  Month 6: number analyzed (Participants) | 52
  Month 6 | 0
  Month 8: number analyzed (Participants) | 48
  Month 8 | 0
  Month 10: number analyzed (Participants) | 42
  Month 10 | 0
  Month 12: number analyzed (Participants) | 40
  Month 12 | 0
  Month 18: number analyzed (Participants) | 26
  Month 18 | 0
  Month 24: number analyzed (Participants) | 23
  Month 24 | 0
  Month 30: number analyzed (Participants) | 10
  Month 30 | 0
  Month 36: number analyzed (Participants) | 8
  Month 36 | 0
  Month 42: number analyzed (Participants) | 1
  Month 42 | 0

24. Secondary Outcome: Ratio of Afatinib Tablets Actually Taken to Doses Prescribed Over the Study Participation Period
Description: Ratio of afatinib tablets actually taken to doses prescribed over the study participation period. Ratio = doses taken / doses prescribed.
Time Frame: Up to 42 months.
Population: All eligible subjects who have been enrolled into the study regardless of whether or not they have finally completed their projected participation in the study and who were evaluable for treatment adherence.
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 63
Ratio | 0.99 (0.02)

25. Secondary Outcome: Number of Patients With a Reason for Missing Afatinib Tablets
Description: Number of patients with a reason for missing afatinib tablets. One participant can have multiple missing doses for multiple reasons.
Time Frame: Up to 42 months.
Population: All subjects who were evaluable for treatment adherence and had missed doses. One participant can have multiple missing doses for multiple reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 11
Participants
  Patients' initiative due to adverse event | 11
  Patient's negligence | 1
  Travel | 1

26. Secondary Outcome: Number of Patients With a Reason for Discontinuation of Afatinib
Description: Number of patients with a reason for discontinuation of Afatinib throughout the study observation period.
Time Frame: Up to 42 months.
Population: All eligible subjects who have been enrolled into the study regardless of whether or not they have finally completed their projected participation in the study and who discontinued treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 56
Participants
  Adverse event | 7
  Disease progression | 43
  Lost to follow-up | 4
  Patient's non-compliance | 1
  Physician's decision | 1

27. Secondary Outcome: Number of Patients With a Reason for Treatment Interruptions
Description: Number of patients with a reason for treatment interruptions throughout the study observation period. One participant can have multiple interruptions for multiple reasons.
Time Frame: Up to 42 months.
Population: All eligible subjects who have been enrolled into the study regardless of whether or not they have finally completed their projected participation in the study and who had treatment interruptions. One participant can have multiple interruptions for multiple reasons.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 26
Participants
  Adverse event/Disease progression | 24
  Physician's advice due to receipt of antibiotic therapy | 2
  Surgery | 2
  Travel | 1
  Physician's decision while waiting for the liquid biopsy results | 1
  Scheduled dental work | 1

28. Secondary Outcome: Number of Participants With Afatinib Interruptions or Dose Modifications
Description: Number of participants with Afatinib interruptions or dose modifications (i.e., a dose increase or decrease).
Time Frame: Up to 42 months.
Population: All eligible subjects that have received at least one dose of Afatinib in the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 77
Participants
  No interruptions/dosage modifications | 42
  Interruptions & Dosage modifications | 17
  Dosage modifications only | 9
  Interruptions only | 9

29. Secondary Outcome: Number of Patients With a Reason for Dose Reduction
Description: Number of patients with a reason for dose reduction throughout the study observation period.
Time Frame: Up to 42 months.
Population: All eligible subjects who have been enrolled into the study regardless of whether or not they have finally completed their projected participation in the study and who had a dose reduction.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 26
Participants
  Adverse event/Disease progression | 23
  Physician's decision (with no further specification) | 1
  Physician's decision due to patient's impaired general health state | 1
  Physician's decision due to patient's impaired performance status | 1

30. Secondary Outcome: Number of Patients With a Reason for Dose Increase
Description: Number of patients with a reason for dose increase throughout the study observation period.
Time Frame: Up to 42 months.
Population: All eligible subjects who have been enrolled into the study regardless of whether or not they have finally completed their projected participation in the study and who had a dose increase.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
Number analyzed (Participants) | 3
Participants
  Physician's decision (with no further specification) | 2
  Adverse event resolution | 1

ADVERSE EVENTS:
Time Frame: Each participant was treated with afatinib and observed in the context of the study until the end of study participation, up to 42 months.
Description: Sufficient data is available to support the evidence on the safety of the studied drug. For this reason, only the following Adverse events of interest were collected and reported:
  * all Adverse Drug Reactions (ADRs),
  * all AEs with fatal outcome,
  * all AEs which were relevant for a serious ADR or an AE with fatal outcome.
  Mortality reporting: all enrolled subjects AE reporting: all eligible enrolled subjects
Arm/Group | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib
All-Cause Mortality (participants affected / at risk) | 7/80
Serious Adverse Events (participants affected / at risk) | 49/77
Other Adverse Events (participants affected / at risk) | 56/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib (N=77)
Anaemia (Blood and lymphatic system disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 1
Death (General disorders) | 2
Pyrexia (General disorders) | 1
Lung abscess (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 45
Dementia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 2
Renal failure (Renal and urinary disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Non-small Cell Lung Cancer (NSCLC) Treated With Afatinib (N=77)
Diarrhoea (Gastrointestinal disorders) | 50
Fatigue (General disorders) | 5
Mucosal inflammation (General disorders) | 5
Conjunctivitis (Infections and infestations) | 6
Paronychia (Infections and infestations) | 15
Decreased appetite (Metabolism and nutrition disorders) | 5
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Dermatitis (Skin and subcutaneous tissue disorders) | 5
Dry skin (Skin and subcutaneous tissue disorders) | 5
Nail dystrophy (Skin and subcutaneous tissue disorders) | 6
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 34
Xeroderma (Skin and subcutaneous tissue disorders) | 4

LIMITATIONS AND CAVEATS:
Main limitations are attributed to its observational design and mainly involve patient selection bias, information bias and missing data as well as lack of internal validity (no control group). Another factor that may have affected Patient Reported Outcomes was the COVID-19 pandemic, which started shortly after the last patient completed their first visit (18 February 2020) thus spanning one out of the total of five years of the study (last patient last visit: 17 February 2021).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2018-07-31): https://cdn.clinicaltrials.gov/large-docs/54/NCT02440854/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02440854/SAP_001.pdf